CLINICAL TRIAL: NCT07102394
Title: Feasibility and Tolerability of IMLYGIC for the Treatment of Cutaneous Neurofibromas in Adults With NF1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Neurofibromatosis Therapeutic Acceleration Program (Unknown); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00482551
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: NF1; Neurofibromatosis; Cutaneous Neurofibroma; Neurofibroma; Von Recklinghausen Disease; Neurofibromas
Keywords: NF1; neurofibromatosis; cutaneous neurofibroma; IMLYGIC; T-VEC; Neurofibromatosis type 1; neurofibroma
MeSH Terms: conditions — Neurofibromatoses; Neurofibroma; Neurofibromatosis 1 | interventions — talimogene laherparepvec

STUDY DESIGN:
Intervention Model Description: This is a single institutional phase 1 study with a safety feasibility and tolerability study of IMLYGIC monotherapy in adults with NF1 and cNFs in need of treatment. Each 28-day treatment cycle will be defined as intralesional administration of IMLYGIC administered on Days 1 and 21 of each cycle for 4 cycles (8 treatments).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMLYGIC (Experimental): 28-day treatment cycle will be defined as intralesional administration of IMLYGIC administered on Days 1 and 21 of each cycle for 4 cycles (8 treatments).
  Interventions: Drug: Imlygic

INTERVENTIONS:
Drug: Imlygic — intralesional administration of IMLYGIC administered on Days 1 and 21 of each cycle for 4 cycles (8 treatments).

SUMMARY:
This study is designed to establish the foundation for a new therapy for neurofibromatosis Type I (NF1)-related cutaneous neurofibromas (cNFs) by assessing the feasibility and efficacy of IMLYGIC in adults with NF1 and cNFs who desire local treatment of their cNF due to disfigurement, progression, pain, itching or other concerns. This is a single institutional Phase 1 study with a safety run-in to assess the feasibility and efficacy of IMLYGIC monotherapy in NF1 patients with cNFs. Each 28-day treatment cycle will be defined as intralesional administration of IMLYGIC administered on day 1 and 21 of Cycle 1 and days 7 and 21 for Cycles 2-4 for up to 4 cycles.

DETAILED DESCRIPTION:
This is a single institutional feasibility and tolerability study of IMLYGIC monotherapy in adults with NF1 and cNFs in need of treatment. Each 28-day treatment cycle will be defined as intralesional administration of IMLYGIC administered on day 1 and 21 of Cycle 1 and days 7 and 21 for Cycles 2-4 for up to 4 cycles. (8 treatments). All patients must be at least 18 years of age or older with at least 8 cNFs measuring 5 mm at minimum in longest diameter, Karnofsky performance status of 80% or higher, and have adequate hematologic, renal and hepatic function. After providing written informed consent to participate in the study, patients will be evaluated for study eligibility during the screening visits.

During screening, a complete medical history will be documented, and a complete physical examination will be conducted. Measurement of vital signs and Karnofsky performance status will be obtained. Laboratory samples will be collected to assess hematologic, renal, and hepatic function. The investigators will also collect a sample to evaluate Herpes Simplex-1 (HSV1) DNA Polymerase Chain Reaction (PCR), HSV1 Immunoglobin G (IgG) and Immunoglobin M (IgM) antibodies, these will be Clinical Laboratory Improvement Amendments (CLIA) certified laboratory tests at baseline and at the end of the study. Patients should be treated until week 16 (4 months). After 16 weeks, patients will remain on study for 30-days to allow post-treatment assessment. If a participant achieves a complete response (cutaneous neurofibromas resolve and are no longer visible) for all of the target tumors before the end of the planned treatment, then the study drug will be stopped at that point, but the patient will be seen at the 30 day mark post last treatment in all cases. Efficacy assessment will be based on tumor measurement by physical measurement, photographs of superficial lesions, and representative biopsy of residual masses suspected. After cycles 2, 4 and at End of Treatment (EOT), a thorough assessment of the clinical response status will be made, particularly to determine if any evidence of biological activity of treatment can be observed.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age ≥ 18 years who meet the NIH clinical criteria for the diagnosis of NF1
* Must have ≥8 measureable cNFs. Histologic confirmation of tumor is not necessary in the presence of consistent clinical findings or confirmed genetic testing. A Measurable cNF is defined as a cutaneous lesion that meets these criteria:
* Singular lesion surrounded by uninvolved skin measuring ≥ 5 mm in the longest diameter but not larger than 5 cm

  1. Not covered by hair
  2. There is no skin breakdown in the tumor or the skin around it
  3. Not located in an area that is prone to irritation or trauma.
  4. A tumor that has not received other therapies such as electrodessication, laser treatment, or prior resection or biopsy.
  5. Diffusely infiltrating cutaneous neurofibromas, subcutaneous neurofibromas, and plexiform neurofibromas are NOT eligible for treatment as photographic assessments and measurements with calipers or ruler are not possible or reliable.
  6. Participants must have 6 cNFs that are amenable for excision.
  7. Participants must be willing to undergo pre- and post-treatment tumor excisions providing fresh tumor tissue; there should be no contraindication for serial biopsies.
* Karnofsky performance level of ≥ 80%.
* Adequate organ and bone marrow and other organ function as defined by the following Screening laboratory values:

  1. Absolute neutrophil count ≥ 1,500 cells/µL;
  2. Platelets ≥ 100 x 103/µL;
  3. Hemoglobin ≥ 9.5 g/dL;
  4. Serum albumin ≥ 2.8 g/dL;
  5. Calculated creatinine clearance at Screening ≥ 60 mL/min (by Cockcroft-Gault formula) OR a normal serum creatinine.
  6. Alanine aminotransferase (ALT) ≤ 2x upper limit of institutional norm
  7. Total bilirubin value of ≤1.5 x Upper Limit of Normal (ULN) (isolated bilirubin ≥1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Participant is willing and able to comply with all aspects of the protocol
* Ability to understand and willingness to sign written informed consent document(s).
* Women of childbearing potential (WOCBP) must not be pregnant or breastfeeding during any portion of the study and must use an adequate method to prevent pregnancy during the study period and for 3 months after treatment conclusion and agree not to donate eggs (ova, oocytes) for the purpose of reproduction during the study and for a period of 3 months after last dose of study treatment. The Investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study treatment (see the Approved Methods of birth control listed below).
* For a woman to be determined not of childbearing potential, she must have ≥ 12 months of non-therapy-induced amenorrhea or be surgically or medically sterile.
* WOCBP must have a negative serum pregnancy test result at Screening and a negative urine pregnancy test result at the Baseline visit prior to the first dose of study treatment if the Screening Day serum test was done more than 28 days prior.
* Male participants are eligible to participate if agreed to the following during the treatment period and for at least 90 days after the last dose of study treatment:

  -- Refrain from donating sperm
* PLUS, either:

  * Be abstinent from heterosexual intercourse and agree to remain abstinent until 90 days after the last study drug treatment; OR
  * Must agree to use a male condom when having sexual intercourse with a WOCBP and their female partner must utilize one the approved methods of birth control below:
* Approved Methods of birth control for this study are:

  * Total abstinence
  * Male or female sterilization (vasectomy in males or surgical removal of ovaries or uterus in females)
  * Unsterilized male study participants must use a male condom, and their female partner must use one of the methods below:
  * Unsterilized female study participants must use one of the following highly effective methods listed below:
* Acceptable birth control methods which are considered highly effective if methods result in a failure rate of less than 1% per year when used consistently and correctly:
* Combined (estrogen and progestogen containing) hormonal contraceptive that stops the release of eggs from the ovary (oral, intravaginal, or transdermal)
* Progestogen-only hormonal contraception that stops the release of eggs from the ovary (oral, injectable, implantable)
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion or bilateral tubal ligation

Exclusion Criteria:

* Any underlying medical condition, which in the opinion of the investigator, would make administration of the study drug hazardous or make it difficult to monitor adverse effects.
* Evidence of immunosuppression for any reason:

  1. Known HIV infection or AIDS
  2. Acute or chronic active hepatitis B or hepatitis C infection
  3. Chronic oral or systemic steroid medication use at a dose of >10 mg/day of prednisone or equivalent (steroids with low systemic absorption [e.g., triamcinolone hexacetonide] is allowed)
  4. Other signs or symptoms of clinical immune system suppression
* Open herpetic skin lesions
* Any anti-herpetic treatment within the last 4 weeks prior to trial participation
* Require intermittent or chronic treatment with an anti-herpetic drug (e.g., acyclovir, valacyclovir, famciclovir, any other antiviral medications), other than intermittent topical use
* One year since the last treatment for any cancer, and not requiring any ongoing secondary prevention, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Patients who have had chemotherapy or radiation therapy must have recovered normal organ function as defined above; people who had excisions of basal cell or squamous cell carcinoma, must have healed and the scars must be at least 3 cm away from any cNF being monitored or treated.
* Active optic glioma or other low-grade glioma or plexiform neurofibroma requiring treatment. a. Participants not requiring treatment are eligible.
* Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) or long-standing orbito-temporal Plexiform Neurofibroma (PN) (such as visual loss, strabismus) are eligible
* Patients with marked baseline prolongation of QT/QTc interval (QTc interval >470 msec) must be excluded.
* Previous treatment with IMLYGIC or treatment with Granulocyte-macrophage colony-stimulating factor (GM-CSF)
* Currently receiving therapy with a Mitogen-Activated Protein Kinase (MEK) inhibitor or treated with a MEK inhibitor in the 6 months prior to the first dose of study treatment.
* Pregnant or breastfeeding women may not take study drug.
* Current enrollment or past participation in any other clinical study (excluding observational studies) within 30 days of the first dose of study treatment.
* Known sensitivity to the study treatment, or components thereof, or drug or other allergy that, could compromise safety of the subject
* Participants are excluded if they have severe and/or uncontrolled medical disease or social situation, which could compromise participation in the study (e.g., uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration, congestive heart failure, drug or alcohol dependence, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of IMLYGIC as assessed by percentage of participants receiving 4 treatments | 1 year
  Feasibility is defined as ≥80% of participants receiving 4 treatments
Tolerability of IMLYGIC as assessed by participants without Dose Limiting Toxicity (DLT) or Serious Adverse Event (SAE) | 1 year
  Tolerability is defined as no participants have a DLT or SAE

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Romo, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States